CLINICAL TRIAL: NCT04762394
Title: Epidemiology of Psychiatric Disorders Among Preschool and School Children and Adolescent in Egypt
Brief Title: Epidemiology of Psychiatric Disorders in Children and Adolescent at Egypt
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Gellan Karamalllah Ramadan Ahmed, lecturer, resarcher OF Neurology and Psychiatry department, Assiut University
Other Study IDs: Assiut university, Egypt
Record Dates: First submitted 2021-02-15; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Child Behavior Disorders; Child Mental Disorder; Adolescent Behaviour Disorder
Keywords: child; adolescent; psychiatry
MeSH Terms: conditions — Child Behavior Disorders; Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: The Child Behavior Checklist (CBCL), — It consists of 113 items; the parents complete it to detect emotional and behavioural problems in children and adolescents aged 6 to 18 years. It is scored on a three-point Likert scale (0=absent, 1= occurs sometimes, 2=occurs often). The time duration for item responses is the past six months.

SUMMARY:
Pediatric, developmental and mental health problems are more common than renal, cardiac and renal problems.

Compartmental problems were often conceptualised across two broad spectrums: internalising intrapersonal problems like anxiety, depression and withdrawal and externalising problems such as Interpersonal problems such as hyperactivity and aggression.

Mental disorders with long-term consequences can result in children and adolescents, undermining health compliance and reducing societies' ability to be safe and productive. As, children and adolescent have long-term deteriorating effects of mental health problems are often serious.

Early detection and identification of problems are in the best interest of children, adolescents, their families, and the community as a whole. All three are important.

how epidemiology can help our understanding of children and adolescent mental health: the burden of the community, measurement and tracking highly significant.

This study will display the first large-scale study of psychiatric disorders in children and adolescents in the Egypt . to provide services, including prevention and intervention based on evidence of mental health, a population-representative child survey and adolescent mental estimates disorders were needed urgently

ELIGIBILITY:
Inclusion Criteria:

1. age of children (2-18 years)
2. both males and females.
3. living in Egypt.

Exclusion Criteria:

* unwilling parent to recruited in the study.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This is study will take part in community study( nursery and schools).
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-02-20 (Estimated); Primary Completion 2022-02-20 (Estimated); Study Completion 2023-02-20 (Estimated)

PRIMARY OUTCOMES:
measure the prevalence of DSM 5 psychiatric disorders in the community sample of school children in Assiut government. | through study completion, an average of 1 year
  by using The Child Behavior Checklist (CBCL):It consists of 113 items, the parents complete it to detect emotional and behavioural problems in children and adolescents .It includes open-ended items covering physical problems, concerns, and strengths. The CBCL/6-18 yields scores on internalizing, externalizing, and total problems as well as scores on DSM-5 related scales.It is providing a total behaviour problem score and two second order factor scores for internalizing problems (anxious/depressed, somatic complaints, withdrawn/depressed) and externalizing behaviour (rule breaking behaviour and aggressive problems).
measure of risk factor of DSM 5 psychiatric disorders in the community sample of school children in Assiut government. | through study completion, an average of 1 year
  Patients were subjected to a full psychiatric and medical assessment at the beginning of the study. A semistructured form was prepared by researchers to detect sociodemographic and clinical variables of the patients, and the medical history of the patients were reviewed. Information gathered included age, sex, birth order, pregnancy problems, delivery type, birth complications, delay of speech development, delay of motor development, family history of consanguinity

CONTACTS AND LOCATIONS:
Locations (1):
- gellan Ahmed, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No